CLINICAL TRIAL: NCT03041610
Title: Effect of Pedometer-Based Walking Intervention on Functional Capacity and Neurohumoral Modulation in Patients With Chronic Heart Failure With Reduced Ejection Fraction: a Multicenter Randomized Controlled Trial
Brief Title: Pedometer-Based Walking Intervention in Patients With Chronic Heart Failure With Reduced Ejection Fraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charles University, Czech Republic (Other)
Collaborators: University Hospital Hradec Kralove (Other); University Hospital Olomouc (Other); Tomas Bata Hospital, Czech Republic (Other); Brno University Hospital (Other); General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Jan Belohlavek, Ass. Prof., Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Walking in HFrEF
Record Dates: First submitted 2017-01-29; First posted 2017-02-03 (Estimated); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Systolic Heart Failure
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walking intervention (Experimental)
  Interventions: Behavioral: Walking intervention
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Walking intervention — The intervention will be delivered over a six-month period and will consist of: (1) an individualized pedometer-based walking program with weekly step goals, (2) regular visits to the clinic including face-to-face session with the physician, and (3) regular telephone calls with the research nurse in between the face-to-face contacts.
  Arms: Walking intervention

SUMMARY:
A multicenter randomized controlled trial, with follow-up at 6 and 12 months. Physically inactive participants with chronic heart failure with reduced ejection fraction will be randomly assigned to intervention or control arms.

The six-month intervention will consist of an individualized pedometer-based walking program with weekly step goals, monthly face-to-face sessions with the physician, and monthly telephone calls with the research nurse. The intervention will be based on effective behavioral principles (goal setting, self-monitoring, personalized feedback).

The primary outcome is the change in 6-minute walk distance at 6 months. Secondary outcomes include changes in serum biomarkers levels, pulmonary congestion assessed by ultrasound, average daily step count measured by accelerometry, anthropometric measures, symptoms of depression, health-related quality of life, self-efficacy, and MAGGIC Risk Score.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of heart failure with reduced ejection fraction (left ventricular ejection fraction <40%) with New York Heart Association (NYHA) class II or III symptoms.
2. Physically inactive, as determined by a question "As a rule, do you do at least half an hour of moderate or vigorous exercise (such as walking or a sport) on five or more days of the week?".

Exclusion Criteria:

1. Signs and symptoms of decompensated heart failure, uncontrolled arrhythmia or effort angina, severe or symptomatic aortic stenosis, persistent hypotension, recent shocks delivered by the automated implantable cardioverter defibrillator.
2. Co-morbid conditions that would affect adherence to trial procedures (e.g. inflammatory arthritis, active malignancy, renal disease requiring dialysis, uncontrolled diabetes, major depression or other significant psychiatric disorders, cognitive impairment, significant hearing or visual impairment).
3. Major surgery planned within the next 12 months.
4. Life expectancy shorter than 12 months.
5. Inability to walk from any reason.
6. Baseline six-minute walking distance >450 meters. Patients covering more than 450 meters in the baseline six-minute walk test (6MWT) are excluded due to a possible ceiling effect.
7. Pregnancy.
8. Failure to perform the 6MWT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
functional capacity | 6 months
  functional capacity change measured with 6-minute walk test

SECONDARY OUTCOMES:
functional capacity | 12 months
  functional capacity change measured with 6-minute walk test
NT-proBNP | 6 months
  N-terminal pro-B-type natriuretic peptide levels
hsCRP | 6 months
  high-sensitivity C-reactive protein
pulmonary congestion | 6 and 12 months
  assessed by ultrasound detection of B-lines
physical activity | 6 and 12 months
  average daily step count measured over 7 days by ActiGraph
depression | 6 and 12 months
  assessed with the Beck Depression Inventory-II
health-related quality of life | 6 and 12 months
  assessed with the 36-Item Short Form Health Survey (SF-36)
self-efficacy | 6 and 12 months
  assessed with the Czech version of the General Self-Efficacy scale (DOVE)
body mass index | 6 and 12 months
  calculated by dividing the body weight (kg) by the square of the height (m2).
waist circumference | 6 and 12 months
  recorded with a measurement tape to the nearest 0.1 cm
hip circumference | 6 and 12 months
  recorded with a measurement tape to the nearest 0.1 cm
Meta-Analysis Global Group in Chronic Heart Failure (MAGGIC) Risk Score | 6 and 12 months
  method to predict survival in heart failure patients

CONTACTS AND LOCATIONS:
Overall Officials: Jan Belohlavek, Ass. Prof., Principal Investigator — Charles University, Czech Republic
Locations (1):
- General University Hospital in Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vetrovsky T, Siranec M, Frybova T, Gant I, Svobodova I, Linhart A, Parenica J, Miklikova M, Sujakova L, Pospisil D, Pelouch R, Odrazkova D, Parizek P, Precek J, Hutyra M, Taborsky M, Vesely J, Griva M, Semerad M, Bunc V, Hrabcova K, Vojkuvkova A, Svoboda M, Belohlavek J; WATCHFUL Investigators. Lifestyle Walking Intervention for Patients With Heart Failure With Reduced Ejection Fraction: The WATCHFUL Trial. Circulation. 2024 Jan 16;149(3):177-188. doi: 10.1161/CIRCULATIONAHA.123.067395. Epub 2023 Nov 13. PMID 37955615
- [Derived] Vetrovsky T, Siranec M, Frybova T, Gant I, Semerad M, Miklikova M, Bunc V, Vesely J, Stastny J, Griva M, Precek J, Pelouch R, Parenica J, Jarkovsky J, Belohlavek J. Statistical analysis plan for a randomized controlled trial examining pedometer-based walking intervention in patients with heart failure with reduced ejection fraction: the WATCHFUL trial. Trials. 2023 Aug 17;24(1):539. doi: 10.1186/s13063-023-07516-5. PMID 37587489
- [Derived] Vetrovsky T, Siranec M, Parenica J, Griva M, Stastny J, Precek J, Pelouch R, Bunc V, Linhart A, Belohlavek J. Effect of a 6-month pedometer-based walking intervention on functional capacity in patients with chronic heart failure with reduced (HFrEF) and with preserved (HFpEF) ejection fraction: study protocol for two multicenter randomized controlled trials. J Transl Med. 2017 Jul 3;15(1):153. doi: 10.1186/s12967-017-1257-x. PMID 28673328